CLINICAL TRIAL: NCT04578366
Title: Effects Of Extracorporeal Shockwave Therapy in Long-term Functional Outcomes of Shoulder Adhesive Capsulitis
Brief Title: Extracorporeal Shockwave Therapy in Long-term Functional Outcomes of Shoulder Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RE-MS-OMPT/Spring19/032 Adnan
Record Dates: First submitted 2020-09-25; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwavetherapy Group/Experimental group (Experimental): ESWT along with conventional therapy ESWT + hot pack(10min), ultrasound (5min), mobilizations, stretching, pendulum exercises, isometrics of shoulder
  Interventions: Device: Extracorporeal Shockwave Therapy
- Conventional Group (Active Comparator): Conventional therapy hot pack(10min), ultrasound (5min), mobilizations, stretching, pendulum exercises, isometrics of shoulder
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy — ESWT along with conventional therapy ESWT + hot pack(10min), ultrasound (5min), mobilizations, stretching, pendulum exercises, isometrics of shoulder
  Other Names: Experimental Group
  Arms: Shockwavetherapy Group/Experimental group
Other: Conventional Treatment — hot pack(10min), ultrasound (5min), mobilizations, stretching, pendulum exercises, isometrics of shoulder
  Arms: Conventional Group

SUMMARY:
Adhesive capsulitis refers to the occurrence of pain and a gradual decline in the range of motion (ROM) due to slow increases in synovial hypertrophy and the adhesion between the synovial membrane and articular surface. It leads to the loss of flexibility and difficulties with the activities of daily living (ADLs) due to chronic inflammation accompanied by intra-articular fibrosis. The real cause of this syndrome is unknown but there are some predisposing factors involved such as synovial cell hyperplasia, fibrosis of the capsule due to cytokines or other inflammatory factors. In the current study investigator will compare the effects of Extracorporeal Shockwave Therapy (ESWT) along with conventional therapy to treat the adhesive capsulitis.

DETAILED DESCRIPTION:
This study will be a Randomized Controlled Trail conducted at Horizon hospital, Lahore. The study will be completed within the time duration of Six months. Consecutive sampling technique will be used to collect the data. The sample size of 44 patients will be taken in this study to find the effects of ESWT on pain, ROM, functional mobility. Patient will be divided into two groups. Group A will be treated with ESWT with conventional therapy and Group B will be treated with conventional therapy. Constant Shoulder Score (CSS) and the Oxford Shoulder Score (OSS) tools will be used to measure the outcomes of the study.

One session of treatment per week for four weeks will be given. Pretest, posttest at 4th week and followup of 24th weeks will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or episode of pain score ≥5 at assessment with a past history of pain for at least 2 months.
* ROM restriction (>75% ROM loss in ≥2 directions including abduction, flexion and external rotation)
* No treatment other than analgesics with unresponsive ROM restriction for the past 2months.
* Unwilling or waiting and did not undergo joint injection.

Exclusion Criteria:

* bilateral shoulder involvement
* History of previous surgery on the shoulder
* Shoulder fracture
* Cancer
* Glenohumeral or Acromioclavicular arthritis
* Inflammatory disorders
* Bleeding disorders
* Diabetes mellitus
* Presence of severe osteoporosis
* Pulmonary diseases
* Any neuromuscular disorders
* Pregnancy
* Implanted pacemaker

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Constant Shoulder Score (CSS) | 8 months
  The functional outcome of shoulder. Grading the Constant Shoulder Score (Difference between normal and Abnormal Side)
  >30 Poor 21-30 Fair 11-20 Good <11 Excellent
Range of motion | 8 months
  Oxford Shoulder Score (OSS), increasing score shows improvement, decrease in scores shows deterioration.

SECONDARY OUTCOMES:
NPRS-numeric pain rating scale | 8 months
  This scale ranges 0-10, 10 means severe pain while 0 means no pain

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calis M, Demir H, Ulker S, Kirnap M, Duygulu F, Calis HT. Is intraarticular sodium hyaluronate injection an alternative treatment in patients with adhesive capsulitis? Rheumatol Int. 2006 Apr;26(6):536-40. doi: 10.1007/s00296-005-0022-2. Epub 2005 Aug 10. PMID 16091920
- [Background] Hussein AZ, Donatelli RA. The efficacy of radial extracorporeal shockwave therapy in shoulder adhesive capsulitis: a prospective, randomised, double-blind, placebo-controlled, clinical study. European Journal of Physiotherapy. 2015;18(1):63-76.
- [Background] Massoud SN, Pearse EO, Levy O, Copeland SA. Operative management of the frozen shoulder in patients with diabetes. J Shoulder Elbow Surg. 2002 Nov-Dec;11(6):609-13. doi: 10.1067/mse.2002.127301. PMID 12469088
- [Background] Wohlgethan JR. Frozen shoulder in hyperthyroidism. Arthritis Rheum. 1987 Aug;30(8):936-9. doi: 10.1002/art.1780300815. PMID 3498494
- [Background] Lee S, Lee S, Jeong M, Oh H, Lee K. The effects of extracorporeal shock wave therapy on pain and range of motion in patients with adhesive capsulitis. J Phys Ther Sci. 2017 Nov;29(11):1907-1909. doi: 10.1589/jpts.29.1907. Epub 2017 Nov 24. PMID 29200621
- [Background] Santoboni F, Balducci S, D'Errico V, Haxhi J, Vetrano M, Piccinini G, Ferretti A, Pugliese G, Vulpiani MC. Extracorporeal Shockwave Therapy Improves Functional Outcomes of Adhesive Capsulitis of the Shoulder in Patients With Diabetes. Diabetes Care. 2017 Feb;40(2):e12-e13. doi: 10.2337/dc16-2063. Epub 2016 Nov 29. No abstract available. PMID 27899492
- [Background] Chen CY, Hu CC, Weng PW, Huang YM, Chiang CJ, Chen CH, Tsuang YH, Yang RS, Sun JS, Cheng CK. Extracorporeal shockwave therapy improves short-term functional outcomes of shoulder adhesive capsulitis. J Shoulder Elbow Surg. 2014 Dec;23(12):1843-1851. doi: 10.1016/j.jse.2014.08.010. PMID 25441567